CLINICAL TRIAL: NCT02563756
Title: Unicondylar - or Total Knee Replacement in Medial Gonarthritis? A Randomized Study of Patient Related Outcome Measures, Function and Muscle Mass
Brief Title: Unicondylar- or Total Knee Replacement? Patient Satisfaction, Function and Muscle Mass
Acronym: UKA or TKA?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Margareta Hedström, MD PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UNITKAstudien2015
Record Dates: First submitted 2015-09-18; First posted 2015-09-30 (Estimated); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Knee Osteoarthritis
Keywords: Medial gonarthritis, knee osteoarthritis,; Muscle function, muscle mass, muscle atrophy; Total knee arthroplasty (TKA); Unicondylar knee arthroplasty (UKA); Total knee replacement (TKR); Unicondylar knee replacement (UKR); Health-related quality of life (HRQoL); Patient related outcome measurements (PROMs)
MeSH Terms: conditions — Osteoarthritis, Knee; Muscular Atrophy | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- UKA, unicompartmental knee replacement (Experimental): Procedure: Participants are operated with a mobile bearing medial unicompartmental knee arthroplasty (Oxford). They are followed with CT, functional tests and PROM, compared with those operated with TKA.
  Interventions: Procedure: Unicompartmental knee replacement
- TKA, total knee replacement (Experimental): Procedure: Participants are operated with a cruciate retaining conventional tricompartmental prosthesis (PFC). They are followed with CT, functional tests and PROM, compared with those operated with UKA.
  Interventions: Procedure: Total knee replacement

INTERVENTIONS:
Procedure: Unicompartmental knee replacement — Participants with a medial gonarthritis are operated with a medial unicompartmental prosthesis
  Other Names: Oxford
  Arms: UKA, unicompartmental knee replacement
Procedure: Total knee replacement — Participants with a medial gonarthritis are operated with a total knee replacement
  Other Names: PFC
  Arms: TKA, total knee replacement

SUMMARY:
Patients with medial gonarthritis are randomised to a unicompartmental or a total knee replacement.

Primary outcome: Thigh muscle cross sectional area and radiological attenuation measured by CT Secondary aims: functional tests, gait analysis, health related quality of life and patient related outcome.

DETAILED DESCRIPTION:
Objective: The investigators aim with the present study was to compare patient related outcome measurements, knee function and muscle mass in patients operated with an UKR or a TKR for medial gonarthritis.

Hypothesis: The investigators hypothesize that a greater number of patients might benefit from a less invasive surgery in terms of increased quality of life, function and muscle mass.

Primary Outcome: Thigh muscle cross sectional area and radiological attenuation measured by CT.

Secondary outcomes: Functional tests (timed up and go, 30s sit and stand, forward reach, forward step down, 6 min walk and 40 m walk test), knee strength (Biodex isokinetic dynamometer) and patient reported pain on a visual analogue scale (VAS). A number of PROMs: Health related quality of life (EQ-5D), Knee injury and Osteoarthritis Outcome Score (KOOS), Oxford Knee Score (OKS) and Forgotten Joint Score (FJS) as well as 3D movement and gait analysis.

Inclusion criteria: Unilateral medial osteoarthritis of the knee (Kellgren 3b-4), aged 50 or above.

Exclusion criteria: Insufficient anterior cruciate ligament (ACL). Fixed varus deformity >10°, fixed flexion deformity >10°, flexion <100°. Previous high tibial osteotomy on the same side. Any neurological disease affecting strength or locomotion in any leg. Body mass index (BMI) >35. Rheumatoid disease. Symptomatic osteoarthritis of the contra lateral knee or any hip. Insufficient written or spoken Swedish.

ELIGIBILITY:
Inclusion Criteria:

* medial gonarthritis, (Kellgren 3b-4)
* correctible varus deformity less than 10 degrees
* intact ACL
* proficient in written and spoken swedish

Exclusion Criteria:

* Valgus gonarthritis
* flexion deformity of 10 degrees
* knee flexion of less than 100 degrees
* previous high tibial osteotomy
* neuromuscular disorders of lower extremities
* symptomatic osteoarthritis of the contralateral knee or any hip.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Muscle mass | 2 years
  Thigh muscle cross sectional area and radiological attenuation measured by CT

SECONDARY OUTCOMES:
Muscle function | 2 years
  Functional test of quadriceps strength, a stair negotiation test where the patient is asked to perform as many repetitions as possible in 30 seconds.
Health related outcome measurement, questionnaire | 2 years
  EQ5D, a qualitative measurement of patient perceived quality of life
Patient reported outcome measurement, knee function questionnaire (PROM). | 2 years
  Knee osteoarthritis outcome score (KOOS).

CONTACTS AND LOCATIONS:
Overall Officials: Margareta Hedström, MD,PhD, Principal Investigator — CLINTEC, Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden